Official Title: Effect of Tongue-to-Palate Resistance Training on Penetration-

Aspiration Scale and Suprahyoid Muscle Electrical Activity in Geriatric Patients

with Oropharyngeal Dysphagia: A Randomized Control Trial

Kuntjoro Harimurti<sup>1</sup>, Melinda Harini<sup>2</sup>, Bunga Saridewi Nurmansyah<sup>2</sup>, I Wayan Murna

Yonathan<sup>3</sup>, Mohamad Yanuar Amal<sup>3</sup>, Steven Setiono<sup>2</sup>, Boya Nugraha<sup>4</sup>

<sup>1</sup> Department of Internal Medicine, Cipto Mangunkusumo Hospital, University of

Indonesia, Jakarta, Indonesia

<sup>2</sup> Department of Physical Medicine and Rehabilitation, Cipto Mangunkusumo Hospital,

University of Indonesia, Jakarta, Indonesia

<sup>3</sup> Department of Radiology, Cipto Mangunkusumo Hospital, University of Indonesia,

Jakarta, Indonesia

<sup>4</sup> Department Rehabilitation Medicine, Hannover Medical School, Germany

Running Title: TPRT and Swallowing Function in Geriatric Dysphagia

Word counts: 2,927 words

**Number of tables: 5** 

**Number of figures:** 1

Abstract

last updated : August, 1st 2025

Background: Oropharyngeal dysphagia is a prevalent geriatric syndrome associated with malnutrition, aspiration, and increased morbidity. Tongue-to-palate resistance training (TPRT) has emerged as a simple, home-based exercise to strengthen swallowing-related musculature, yet evidence in older adults remains limited.

Objective: This study aimed to evaluate the effects of TPRT on suprahyoid muscle activity and swallowing safety, assessed by the Penetration-Aspiration Scale (PAS), in geriatric patients with oropharyngeal dysphagia.

Methods: A single-blind randomized controlled trial was conducted at Cipto Mangunkusumo Hospital, Jakarta, from July 2022 to June 2024. Twenty patients aged >60 years with videofluoroscopic-confirmed dysphagia were randomized into TPRT and control groups. The intervention group performed TPRT (30 repetitions, five sessions per week, for eight weeks), while controls received individualized dysphagia therapy (neuromuscular electrical stimulation, CTAR, or biofeedback). Suprahyoid muscle activity was measured using surface electromyography (sEMG) at baseline, week 4, and week 8; swallowing function was evaluated using PAS and videofluoroscopic parameters.

Results: Seventeen participants completed the study (intervention n=9, control n=8). Both groups demonstrated significant within-group increases in suprahyoid muscle activity over eight weeks (p<0.001), with larger effect sizes observed in the TPRT group, although between-group differences were not statistically significant. PAS scores improved in both groups [intervention: median  $4\rightarrow2$ ; control:  $4.5\rightarrow2$ ], without significant intergroup differences. Notably, anterior hyoid excursion significantly increased in the TPRT group (p=0.038).

Conclusion: TPRT enhanced suprahyoid muscle activity and anterior hyoid movement in older adults with oropharyngeal dysphagia, supporting its feasibility as a home-based intervention. Although no significant reduction in PAS was observed, TPRT shows promise as a safe, low-cost rehabilitation strategy warranting further investigation in larger, more homogenous cohorts.

# Introduction

Oropharyngeal dysphagia is highly prevalent among older adults, affecting 30–40% of individuals over the age of 65 and over 60% of those in long-term care facilities.<sup>1,2</sup> This condition, characterized by impaired bolus formation and transit from the oral cavity to the esophagus, may lead to aspiration and choking<sup>3,4</sup>, and has been classified as one of the geriatric giants by the European Union Geriatric Medicine Society (EUGMS) and the European Society for Swallowing Disorders (ESSD) due to its impact on nutritional status, functional decline, morbidity, and mortality.<sup>4–6</sup>

Age-related physiological changes, including reduced tongue strength, diminished laryngeal elevation, and weakened suprahyoid muscle activity, contribute to impaired swallowing efficiency. Tongue strength is essential for effective bolus propulsion and generating adequate intraoral pressure, directly influencing the pharyngeal phase of swallowing. Phase of swallowing efficiency, Rehabilitation strategies, such as Shaker or CTAR (Chin Tuck Against Resistance) exercises and neuromuscular electrical stimulation (NMES), are frequently employed but may be unsuitable for frail elderly patients due to physical limitations or low adherence.

Tongue-to-palate resistance training (TPRT), performed by pressing the tongue against the palate, offers a simple and feasible alternative that can be implemented as a home-based program. TPRT has been shown to enhance both anterior and posterior tongue strength, increase hyoid bone excursion, and improve upper esophageal sphincter opening by activating the suprahyoid muscles. 11,14,15

Several studies also report a correlation between tongue movement and suprahyoid muscle activation, with surface electromyography (sEMG) confirming greater suprahyoid activity during TPRT compared to Shaker exercises. 14,16–18

The effects of tongue and suprahyoid muscle strengthening exercises are also supported by findings of increased geniohyoid muscle thickness from 2.3 to 2.6 cm<sup>2</sup> after eight weeks of training,<sup>7</sup> as well as increased thickness of the mylohyoid and digastric muscles following tongue-to-palate pressing exercises performed over six weeks.  $^{9,19}$  A TPRT program consisting of 30 repetitions, five times per week for four weeks, also reduced PAS scores from 6 to 3.56 (p < 0.000).  $^{20}$ 

A preliminary study conducted at the Department of Physical Medicine and Rehabilitation, Cipto Mangunkusumo Hospital, showed an increase in suprahyoid muscle electrical activity from  $8.56\pm3.456~\mu V$  before TPRT to  $15.26\pm3.19~\mu V$  after one week of training, and further increased to  $17.44\pm3.922~\mu V$  after two weeks. <sup>13</sup> Since the strength of both the tongue and suprahyoid muscles can improve solely through tongue-strengthening exercises, TPRT has the potential to enhance swallowing function in both the oral and pharyngeal phases in patients with dysphagia, and may be suitable as a home-based training program. This study aims to evaluate the effect of tongue-to-palate resistance training in geriatric patients with oropharyngeal dysphagia over a longer observation period than typical hospital-based rehabilitation. The outcomes assessed include suprahyoid muscle electrical activity and the Penetration-Aspiration Scale (PAS) to determine the effectiveness of the training and the risk of aspiration.

#### Methods

### Design, population, and setting

This study was an interventional, single-blind, randomized controlled trial (RCT) conducted at the Department of Medical Rehabilitation, Radiology Unit, and Integrated Geriatric Clinic of Dr. Cipto Mangunkusumo General Hospital, Jakarta, between July 2022 and June 2024.

Eligible participants were geriatric patients aged >60 years diagnosed with oropharyngeal dysphagia confirmed through videofluoroscopic swallowing study (VFSS). Inclusion criteria required that participants had not received swallowing training in the preceding two weeks, were cooperative, and had a caregiver available to support adherence to the intervention protocol. Baseline suprahyoid muscle electrical activity, measured by surface electromyography (sEMG), had to be  $\leq$ 37.1  $\mu$ V RMS. Exclusion criteria included significant cognitive impairment based on the MoCA-Ina test, history of radical neck dissection, malignancy of the oral cavity, recent head and neck chemoradiotherapy within three months, complete inability to move the tongue, baseline EMG = 0  $\mu$ V, presence of a pacemaker, or known allergies to contrast agents or training materials.

All participants provided written informed consent prior to enrollment. Ethical approval was obtained from the Research Ethics Committee of the Faculty of Medicine, Universitas Indonesia/Dr. Cipto Mangunkusumo Hospital (No. KET-1415/UN2.F1/ETIK/PPM.00.02/2022)

# Sample Size

The sample size was determined using a paired-mean difference calculation. For suprahyoid muscle electrical activity, the standard deviation of the mean difference was estimated at 3.68 with an expected mean difference of 4.0. Using a significance level of  $\alpha = 0.05$  ( $Z\alpha = 1.96$ ) and power of 80% ( $Z\beta = 0.84$ ), the required minimum sample size was seven subjects.

For the Penetration-Aspiration Scale (PAS), the standard deviation of the mean difference was estimated at 1.03 with an expected mean difference of 1.0, yielding a minimum sample size of eight subjects under the same statistical assumptions. To ensure adequate power, the larger estimate of eight participants per group was selected.

Accounting for an anticipated 20% dropout or loss to follow-up, the final target sample size was set at 20 participants, with 10 allocated to each group.

Baseline measurement, randomization and intervention

Following consent and initial assessments, participants underwent baseline VFSS and suprahyoid sEMG evaluations. Block-permuted randomization with a block size of four was used to allocate subjects into intervention and control groups.

The intervention group received TPRT home exercises consisting of 30 repetitions per session, five sessions per week, over eight weeks with video guidance and support from caregiver. Participants were monitored via logbooks and follow-up calls.

The control group received individualized dysphagia therapy, which may have included neuromuscular electrical stimulation (NMES), biofeedback swallowing therapy, and home-based chin tuck against resistance (CTAR) exercises. NMES

involved placing electrodes in the submental region. Both groups received education on safe swallowing techniques, posture, and bolus modification.

#### Follow-up and outcomes measurement

Suprahyoid sEMG was reassessed at weeks 4 and 8. VFSS parameters (PAS score, pharyngeal transit time, hyoid movement) were evaluated again at week 8. sEMG was recorded using surface electrodes placed in the submental area after skin preparation. Electrode placement was confirmed by asking participants to press their tongue against the palate and perform a dry swallow. Each test was performed three times, with at least 10 seconds of rest between trials to prevent fatigue.

The outcomes measured were suprahyoid muscle electrical activity and the Penetration-Aspiration Scale (PAS).

#### Blinding

Outcome assessors were blinded to group allocation. Suprahyoid muscle electrical activity (sEMG) was evaluated before and after the intervention by a rehabilitation medicine physician, while videofluoroscopic swallowing studies (VFSS) were conducted by a radiologist and a rehabilitation medicine specialist. All assessors were unaware of participants' treatment assignment.

To ensure comparability across groups, both the intervention and control groups also received standard education on posture adjustment, swallowing maneuvers, and bolus modification for safe swallowing.

#### Harms

Adverse events were systematically monitored throughout the study. Participants and caregivers were instructed to report any kejadian tidak diharapkan (adverse events) via telephone during scheduled follow-up logbook checks. This approach ensured continuous surveillance during both the home-based exercise program and the hospital-based assessments. No adverse events were reported in either the intervention or control groups, whether during the training sessions or during outcome evaluations such as suprahyoid sEMG recordings and videofluoroscopic swallowing studies (VFSS) Statistical analysis

Data were presented using narrative summaries and tabular formats. Statistical analysis was conducted using both descriptive and inferential approaches. The normality of EMG data was tested using the Shapiro–Wilk test. If data were not normally distributed, a log transformation was applied. Repeated measures ANOVA (General Linear Model approach) was used to assess time-related effects, with Mauchly's test of sphericity applied to test variance assumptions. If sphericity was violated, corrections (Greenhouse–Geisser or Huynh–Feldt) were applied. For other outcomes, paired t-tests or Wilcoxon signed-rank tests (for within-group comparisons) and independent t-tests or Mann–Whitney U tests (for between-group comparisons) were used based on data distribution. A p-value < 0.05 was considered statistically significant.

#### **Results**

# Recruitment and randomization

A total of 36 patients were screened for eligibility. Sixteen were excluded for the following reasons: suprahyoid EMG activity >37.1  $\mu$ V RMS (n = 3), cognitive impairment (n = 5), history of radical neck dissection (n = 3), pacemaker implantation (n = 2), absence of a consistent caregiver (n = 1), and refusal to participate (n = 2). Twenty eligible participants were randomized using block-permuted randomization with a block size of four, resulting in 10 participants allocated to the intervention group and 10 to the control group. This sample met the minimum number required based on the a priori sample size calculation.

All participants completed the first four weeks of training and underwent the week-4 suprahyoid sEMG assessment. By week 8, three participants withdrew: one from the intervention group due to hospitalization for vascular stenting, and two from the control group (one lost to follow-up and one relocated). In total, 17 participants (intervention n = 9, control n = 8) completed the study and were included in the final analysis. The participant flow and reasons for exclusion and withdrawal are summarized in **Figure 1** (CONSORT flow diagram). The recruitment period spanned from July 2022 to June 2024.

No adverse events were reported during training sessions or during outcome evaluations, including suprahyoid sEMG and VFSS assessments.



**Figure 1.** CONSORT 2010 flow diagram of participant recruitment, randomization, follow-up, and analysis in the TPRT trial

# <u>Intervention and comparator delivery</u>

All participants in the intervention group adhered to the tongue-to-palate resistance training (TPRT) protocol, consisting of 30 repetitions per session, five sessions per week, performed at home with caregiver support, video guidance, and logbook monitoring. In the control group, participants received the standard hospital-based protocol of neuromuscular electrical stimulation (NMES) or biofeedback twice weekly, followed by unsupervised home-based chin-tuck against resistance (CTAR)

exercises. Both groups were able to complete their assigned interventions as scheduled during the study period.

# Concomitant care

Both groups additionally received standardized education on posture adjustment, swallowing maneuvers, and bolus modification to ensure safe swallowing.

# Patients' characteristics

A total of 17 participants completed the full 8-week protocol, including suprahyoid surface electromyography (sEMG) and videofluoroscopic swallowing study (VFSS) assessments. Due to non-normal distribution of sEMG data, natural log transformation was applied, and repeated measures ANOVA (GLM approach) was used for analysis. Baseline characteristics are summarized in Table 1. The mean age of all subjects was  $70.18 \pm 6.24$  years, with no significant age difference between the intervention group ( $69.67 \pm 4.67$  years) and the control group ( $70.75 \pm 7.97$  years). Male participants accounted for 58.8% of the sample, with a slightly higher proportion in the control group (62.5%) than in the intervention group.

Body mass index (BMI) was non-normally distributed and showed no significant difference between groups, with a median of 22.14 (19.22–30.41) kg/m² in the intervention group and 21.14 (16.9–29.4) kg/m² in the control group. The Charlson Comorbidity Index (CCI) was slightly higher in the intervention group [median 6 (3–8)] compared to the control group [median 5 (3–8)]. The proportion of frailty was marginally higher in the control group (62.5%) than in the intervention group (55.6%).

The most common etiology of dysphagia was stroke (47.1%), followed by laryngopharyngeal reflux (LPR, 41.2%) and nasopharyngeal malignancy (11.8%). The baseline PAS score was 4 (2–8) in the intervention group and 4.5 (2–8) in the control group. Penetration (70.6%) was more prevalent than aspiration (29.4%) across both groups.

# Table 1 Patients' characteristics

| | | Group | |
|-------------------|------------------|--------------|-------------|
| Characteristics | Total | Intervention | Control |
| | | (n=9) | (n=8) |
| Age (years) | 70,18 ±6,24 | 69,67 ±4,67 | 70,75 ±7,97 |
| 60-69 | 10 (58,8%) | 6 (66,7%) | 4 (50%) |
| 70-79 | 6 (35,3%) | 3 (33,3%) | 3 (37,5) |
| >80 | 1 (5,9%) | 0 (0%) | 1 (12,5%) |
| Gender | | | |
| Male | 10 (58,8%) | 5 (55,6%) | 5 (62,5%) |
| Female | 7 (41,2%) | 4 (244,4%) | 3 (37,5%) |
| BMI (kg/m²) | 21,6(16,9-30,41) | 22,14(19,22- | 21,14(16,9- |
| | | 30,41) | 29,4) |
| CCI | 5(3-8) | 6(3-8) | 5(3-8) |
| Mild | 0 (0%) | 0 (0%) | 0 (0%) |
| Moderate | 6 (35,3%) | 3 (33,3%) | 3 (37,5%) |
| Severe | 11 (64,7%) | 6 (66,6%) | 5 (62,5%) |
| Frailty | | | |
| Yes | 10 (58,8%) | 5 (55,6%) | 5 (62,5%) |
| No | 7 (41,2%) | 4 (44,4%) | 3 (37,5%) |
| Etiology | | | |
| Stroke | 8 (47,1%) | 4 (44,4%) | 4 (50%) |
| Laryngopharyngeal | 6 (35,3%) | 4 (44,4%) | 2 (25%) |
| Reflux (LPR) | | | |
| Nasopharyngeal | 3 (17,6%) | 1 (11,1%) | 2 (25%) |

#### cancer

| Dysphagia severity | 5(2-8) | 4(2-8) | 4,5(2-8) |
|--------------------|------------|-----------|-----------|
| (PAS) | | | |
| Penetration | 12 (70,6%) | 7 (77,8%) | 5 (62,5%) |
| Aspiration | 5 (29,4%) | 2 (22,2%) | 3 (37,5%) |

# Suprahyoid Muscle Electrical Activity

Baseline measurements showed comparable activity between the intervention and control groups in both tongue-pressed and dry swallowing conditions. At week 4 and week 8, the intervention group showed an increase in median electrical activity during tongue-pressed movements from 34.54 (24.32–36.91) μV RMS to 49.12 (31.28–58.42) μV and 60.87 (28.84–95.79) μV respectively. The control group exhibited a smaller increase from 32.26 (23.42–34.89) μV to 33.13 (30.13–54.38) μV and 42.99 (25.55–89.04) μV. During dry swallowing, the intervention group improved from 35.38 (25.95–36.99) μV RMS at baseline to 50.06 (29.75–69.85) μV at week 4 and 63.91 (27.32–91.99) μVat week 8. The control group increased from 33 (21.43–35.80) μV to 32.14 (24.7–59.15) μV and 54.04 (31.13–85.37) μV. Table 2 describes the increase in suprahyoid muscle electrical activity in both the intervention and control groups during tongue-pressed and dry swallowing movements. Both groups had similar baseline values in tongue-pressed movement as well as in dry swallowing.

**Table 2.** Suprahyoid Muscle Activity Before and After Training in the Intervention and Control Groups

| Suprahyoid muscle | Baseline | Week 4 | Week 8 |
|---|---|---|---|
| electrical activity | | | |
| Tongue pressed (µVF | RMS) | | |
| Intervention | 34,54(24,32-36,91) | 49,12(31,28-58,42) | 60,87(28,84-95,79) |
| Control | 32,26(23,42-34,89) | 33,13(30,13-54,38) | 42,99(25,55-89,04) |
| Dry swallowing (µVF | RMS) | | |
| Intervention | 35,38(25,95-36,99) | 50,06(29,75-69,85) | 63,91(27,32-91,99) |
| Control | 33(21,43-35,80) | 32,14(24,7-59,15) | 54,04(31,13-85,37) |

Repeated Measures ANOVA (GLM approach) was performed after log transformation of non-normally distributed data. Mauchly's test of sphericity indicated violation of the assumption (p < 0.05), requiring Greenhouse-Geisser correction. The results indicated a significant time effect for both tongue-pressed (p = 0.000,  $\eta^2$  = 0.693) and dry swallowing (p = 0.000,  $\eta^2$  = 0.669), while time\*group interaction was not significant, indicating similar patterns of change in both groups. Between-group effects analysis did not yield statistically significant results (p > 0.05), though effect sizes were moderate to large ( $\eta^2$  = 0.164 for tongue pressed,  $\eta^2$  = 0.123 for dry swallow), suggesting a potential clinical impact. Figure 1 illustrates the trend of mean log-transformed suprahyoid muscle activity during tongue-pressed and dry swallowing tasks across baseline, week 4, and week 8, showing a consistent increase in both the intervention and control groups, with greater improvement observed in the intervention group.



Figure 1. General Linear Model of Suprahyoid Muscle Electrical Activity

# Penetration-Aspiration Scale (PAS)

VFSS evaluation prior to the intervention showed similar PAS scores between groups: median (min-max) PAS was 4 (2–8) in the intervention group and 4.5 (2–8) in the control group, with no statistically significant difference (p > 0.05). After completing the training protocol, both groups demonstrated a reduction in PAS at week 8: 2 (1–8) in the intervention group and 2 (1–8) in the control group. However, the difference between groups remained statistically non-significant (p > 0.05). Table 3 presents the comparison of Penetration-Aspiration Scale (PAS) scores between the intervention and control groups at baseline and after 8 weeks of training. While both groups showed a reduction in median PAS scores following the intervention period, no statistically significant differences were observed either within or between groups.

**Table 3.** Comparison of Parameters Before and After Training in the Intervention and Control Groups

| Parameter | Group | Baseline | Week 8 | p-value |
|---|---|---|---|---|
| Anterior hyoid | Intervention | 15.75 (3.21–24.43) | 28.26 (3.5–45.18) | 0.038 <sup>w</sup> |
| mo | | | | |
| ve | | | | |
| me | | | | |
| nt | | | | |
| (% | | | | |
| C2 | | | | |
| _ | | | | |
| C4 | | | | |
| ) | | | | |
| | Control | 14.09 (0.96–17.54) | 14.48 (1.07–23.69) | 0.161 <sup>w</sup> |
| | p-value between groups | $0.178^{\rm m}$ | 0.021 <sup>m</sup> | |
| Superior hyoid | Intervention | 14.52 (5.54–38.85) | 22.07 (4.83–38.33) | $0.086^{w}$ |
| mo | | | | |
| ve | | | | |
| me | | | | |
| nt | | | | |
| (%) | | | | |
| C2 | | | | |
| _ | | | | |
| C4 | | | | |
| ) | | | | |
| | Control | 16.56 (10.68–34.62) | 19.50 (1.77–48.93) | 0.327 <sup>w</sup> |
| | p-value between groups | 0.441 <sup>m</sup> | $0.564^{\rm m}$ | |

| PTT (seconds) | Intervention | 0.63 (0.1–1) | 0.73 (0.23–0.83) | 0.859 <sup>w</sup> |
|---|---|---|---|---|
| | Control | 0.68 (0.5–1) | 0.74 (0.33–5.6) | 0.327 <sup>w</sup> |
| | p-value between groups | 0.923 <sup>m</sup> | $0.310^{\rm m}$ | |
| PAS | Intervention | 4 (2–8) | 2 (1–8) | 0.232 <sup>w</sup> |
| | Control | 4.5 (2–8) | 2 (1–8) | 0.753 <sup>w</sup> |
| | p-value between groups | $1.000^{\rm m}$ | $0.797^{\mathrm{m}}$ | |

# Pharyngeal transit time (PTT)

Other parameters assessed using VFSS in this study included Pharyngeal Transit Time (PTT) and anterior and superior hyoid movement. As shown in Table 3, PTT evaluation revealed no significant differences within or between the intervention and control groups before and after training (p > 0.05).

# Effects of TPRT to hyoid movement

Hyoid movement in the anterior and superior directions was expressed as a percentage of the C2–C4 distance, normalized by dividing each measurement by the length of a straight line connecting the inferior borders of C2 and C4 on the y-axis. Table 3 displays the changes in anterior and superior hyoid excursion. No significant differences were observed between groups at baseline for either direction (p > 0.05). However, in the intervention group, a statistically significant increase was found in anterior hyoid movement between baseline and week 8 (p = 0.038). Additionally, an intergroup comparison at week 8 showed a significant difference in anterior hyoid movement (p = 0.021)

#### **Discussion**

This study aimed to evaluate changes in swallowing function in geriatric patients with oropharyngeal dysphagia by analyzing suprahyoid muscle activity and the Penetration-Aspiration Scale (PAS). Participants were assigned to either a home-based TPRT group using video guidance and logbook monitoring or a control group receiving standard care, including NMES or biofeedback sessions and unsupervised CTAR exercises.

Findings showed that both groups experienced significant increases in suprahyoid muscle activity from baseline to weeks 4 and 8 during tongue-pressed and dry swallowing tasks. While between-group differences were not statistically significant, the large effect sizes observed in the intervention group suggest potential clinical relevance. These results align with previous studies showing improved tongue strength after TPRT or similar resistance training protocols. A more recent study by Kim et al. demonstrated that home-based tongue-to-palate training in stroke patients was as effective as hospital-based programs, with both groups showing significant improvement in tongue muscle strength and volume without differences between the two delivery modes.<sup>41</sup>

Previous studies by Kim et al. reported that the positive effects of TPRT could be observed as early as after 4 weeks of training in tongue muscle strength. <sup>10</sup> Similarly, Plaza et al. found a statistically significant increase in suprahyoid muscle sEMG values by the 4th week of combined tongue-to-palate pressing and strengthening exercises using IOPI, reaching 57.3±13.6 %MVC by the 8th week with tongue-to-palate pressing alone. <sup>21</sup> Resistance training improves muscle performance through neural mechanisms such as increased motor unit recruitment and hypertrophy mediated by muscle IGF and

myogenic factors.<sup>22–24</sup> Robbins et al. further emphasize post-stroke swallowing recovery may involve neuroplasticity.<sup>25–27</sup>

TPRT targets oral and pharyngeal phases of swallowing by strengthening muscles responsible for bolus formation and palatal contact. <sup>15,28,29</sup> The activation of genioglossus and hyoglossus muscles indirectly enhances geniohyoid and suprahyoid activity. <sup>9,17,28,29</sup> Although sEMG reference values vary due to age and normalization methods, a consistent upward trend in sEMG across this study indicates positive training effects. <sup>30–32</sup>

The PAS decreased in both groups by week 8, but without significant between-group differences. Similar findings have been reported in older adults receiving tongue resistance training. <sup>20,33,34</sup> One possible explanation is the "floor effect" in participants with initially low PAS scores, limiting the ability to detect statistical improvements. Additionally, PAS is affected by multiple physiological factors such as pharyngeal timing and hyoid displacement. <sup>35–37</sup> Bingjie et al. identified increased pharyngeal delay time, prolonged pharyngeal transit time, and reduced maximal vertical displacement of the larynx and hyoid bone as independent predictors of aspiration in older adults. <sup>42</sup> Similarly, Zhang et al. demonstrated in a large cohort that anterior hyoid displacement was the most reliable predictor of penetration—aspiration risk, highlighting the critical biomechanical role of hyoid excursion in swallowing safety. <sup>43</sup>

Furthermore, no significant change in PTT was observed, possibly due to participant heterogeneity and age-related physiological changes.<sup>38</sup> In contrast, Namiki et al. reported shortened PTT post-TPRT in a healthier cohort.<sup>11</sup> This study observed statistically significant improvements in anterior hyoid movement among intervention participants. Anterior hyoid displacement is essential for upper esophageal sphincter

(UES) opening and airway protection. Increased anterior hyoid movement suggests neuromuscular adaptations from TPRT, even though PAS scores remained unchanged. These results indicate potential for improving biomechanical aspects of swallowing.<sup>39,40</sup>

In summary, TPRT may enhance suprahyoid muscle activity and anterior hyoid excursion in older adults with oropharyngeal dysphagia. Though PAS and PTT changes were not statistically significant, the observed physiological improvements highlight TPRT as a feasible and promising home-based intervention.

# Strengths and limitations

This is the first randomized controlled trial in Indonesia to evaluate tongue-to-palate resistance training (TPRT) in geriatric patients with oropharyngeal dysphagia. Its simple, equipment-free protocol supports feasibility for home-based use. However, the heterogeneous sample, small sample size, and high data variability may have limited statistical significance despite moderate-to-large effect sizes. A floor effect in PAS scores and use of only thin-liquid consistency for VFSS may also limit generalizability.

# Conclusion

Tongue-to-palate resistance training (TPRT) has the potential to enhance suprahyoid muscle electrical activity in geriatric patients with oropharyngeal phase dysphagia. However, this intervention did not result in a statistically significant reduction in Penetration-Aspiration Scale (PAS) scores in the studied population. This study supports the feasibility of implementing home-based TPRT as a clinical intervention for geriatric patients with oropharyngeal dysphagia. The training protocol may serve as a reference for rehabilitation programs targeting swallowing function in

this population. Future studies should involve larger and more homogenous sample populations to increase statistical power and generalizability. Additionally, longer training durations or combined exercise protocols are recommended to further explore the potential therapeutic effects of TPRT in this patient group.

# **Sources of Funding**

The author did not receive any source of funding.

# **Conflict of Interest**

The author declares no conflict of interest.

#### References

- 1. Clavé P, Rofes L, Carrión S, Ortega O, Cabré M, Serra-Prat M, et al. Pathophysiology, relevance and natural history of oropharyngeal dysphagia among older people. Nestle Nutr Inst Workshop Ser. 2012;72:57–66.
- 2. Clavé P, Rofes L, Arreola V, Almirall J, Cabré M, Campins L, et al. Diagnosis and management of oropharyngeal dysphagia and its nutritional and respiratory complications in the elderly. Gastroenterol Res Pract. 2011;(January).
- 3. Clavé P, Shaker R. Dysphagia: Current reality and scope of the problem. Nat Rev Gastroenterol Hepatol. 2015;12(5):259–70.
- 4. Baijens LWJ, Clavé P, Cras P, Ekberg O, Forster A, Kolb GF, et al. European society for swallowing disorders European union geriatric medicine society white paper: Oropharyngeal dysphagia as a geriatric syndrome. Clin Interv Aging. 2016;11:1403–28.
- 5. Peñalva-Arigita A, Prats R, Lecha M, Sansano A, Vila L. Prevalence of dysphagia in a regional hospital setting: Acute care hospital and a geriatric sociosanitary care hospital: A cross-sectional study. Clin Nutr ESPEN. 2019;33:86–90.
- 6. Smithard DG. Dysphagia: A Geriatric Giant? The Normal Swallow. iMedPub Journals. 2016;2(1:5):1–7.
- 7. Yano J, Yamamoto-Shimizu S, Yokoyama T, Kumakura I, Hanayama K, Tsubahara A. Effects of Tongue-Strengthening Exercise on the Geniohyoid Muscle in Young Healthy Adults. Vol. 35, Dysphagia. 2020. p. 110–6.
- 8. Park T. Effects of Oropharyngeal Strengthening Exercise (OSE) on Tongue Strength, Submental Muscle Activity, and Quality of Life in a Healthy Elderly Population. Ohio University; 2015.
- 9. Park JS, Hwang NK, Kim HH, Choi JB, Chang MY, Jung YJ. Effects of lingual strength training on oropharyngeal muscles in South Korean adults. J Oral Rehabil. 2019;46(11):1036–41.
- 10. Kim HD, Choi JB, Yoo SJ, Chang MY, Lee SW, Park JS. Tongue-to-palate resistance training improves tongue strength and oropharyngeal swallowing function in subacute stroke survivors with dysphagia. J Oral Rehabil. 2017;44(1):59–64.
- 11. Namiki C, Hara K, Tohara H, Kobayashi K, Chantaramanee A, Nakagawa K, et al. Tongue-pressure resistance training improves tongue and suprahyoid muscle functions simultaneously. Clin Interv Aging. 2019;14:601–8.
- 12. Lee KH, Jung ES, Choi YY. Effects of lingual exercises on oral muscle strength and salivary flow rate in elderly adults: a randomized clinical trial. Geriatr Gerontol Int. 2020;20(7):697–703.

- 13. Harini M, Nathania E. The Effectiveness of Tongue Palatal Resistance Training on Increasing Suprahyoid Muscle Strength in Patients with Oropharyngeal Dysphagia: A Home Exercise Program during the Covid-19 Pandemic. ASEAN Journal of Rehabilitation Medicine. 2021;32(Fourthcoming):41–3.
- 14. Reis VS dos, Araújo TG de, Furlan RMMM, Motta AR. Correlation between tongue pressure and electrical activity of the suprahyoid muscles. Revista CEFAC. 2017;19(6):792–800.
- 15. Wirth R, Dziewas R, Beck AM, Clavé P, Hamdy S, Heppner HJ, et al. Oropharyngeal dysphagia in older persons from pathophysiology to adequate intervention: A review and summary of an international expert meeting. Clin Interv Aging. 2016;11:189–208.
- 16. Palmer PM, Luschei ES, Jaffe D, McCulloch TM. Contributions of individual muscles to the submental surface electromyogram during swallowing. Journal of Speech, Language, and Hearing Research. 1999;42(6):1378–91.
- 17. Yoshida M, Groher ME, Crary MA, Mann GC, Akagawa Y. Comparison of surface electromyographic (sEMG) activity of submental muscles between the head lift and tongue press exercises as a therapeutic exercise for pharyngeal dysphagia. Gerodontology. 2007;24(2):111–6.
- 18. Vaiman M. Standardization of surface electromyography utilized to evaluate patients with dysphagia. Head Face Med. 2007;3(1):1–8.
- 19. Park J su, Lee S hoon, Jung S hoon, Choi J bae, Jung Y jin. Tongue strengthening exercise is effective in improving the oropharyngeal muscles associated with swallowing in community-dwelling older adults in South Korea A randomized trial. Medicine. 2019;98(40):1–9.
- 20. Kim HD, Choi JB, Yoo SJ, Chang MY, Lee SW, Park JS. Tongue-to-palate resistance training improves tongue strength and oropharyngeal swallowing function in subacute stroke survivors with dysphagia. J Oral Rehabil. 2017;44(1):59–64.
- 21. Plaza E, Ruviaro Busanello-Stella A. Effects of a tongue training program in Parkinson's disease: Analysis of electrical activity and strength of suprahyoid muscles. Journal of Electromyography and Kinesiology. 2022;63(June 2021):102642.
- 22. Salles B De, Simão R, Fleck S. Effects of Resistance Training on older adults. Sports Medicine. 2010;34(5):441–50.
- 23. Lavin KM, Roberts BM, Fry CS, Moro T, Rasmussen BB, Bamman MM. The importance of resistance exercise training to combat neuromuscular aging. Physiology. 2019;34(2):112–22.
- 24. Gabriel DA, Kamen G, Frost G. Neural adaptations to resistive exercise: Mechanisms and recommendations for training practices. Sports Medicine. 2006;36(2):133–49.
- 25. Robbins JA, Gangnon RE, Theis SM, Kays SA, Hewitt AL, Hind JA. The effects of lingual exercise on swallowing in older adults. J Am Geriatr Soc. 2005;53(9):1483–9.
- Robbins JA, Kays SA, Gangnon RE, Hind JA, Hewitt AL, Gentry LR, et al. The Effects
  of Lingual Exercise in Stroke Patients With Dysphagia. Arch Phys Med Rehabil.
  2007;88(2):150–8.
- 27. Park JS, Kim HJ, Oh DH. Effect of tongue strength training using the iowa oral performance instrument in stroke patients with dysphagia. J Phys Ther Sci. 2015;27(12):3631–4.

- 28. Palmer PM, Jaffe DM, McCulloch TM, Finnegan EM, Van Daele DJ, Luschei ES. Quantitative contributions of the muscles of the tongue, floor-of-mouth, jaw, and velum to tongue-to-palate pressure generation. Dysphagia. 2009;24(1):119.
- 29. Gutierrez DL. A Comparison of Two Devices for Isometric Lingual Strengthening in Healthy Adults A COMPARISON OF TWO DEVICES FOR ISOMETRIC. 2020;(August).
- 30. Furlan R et al. Comparison of the electric activity of the suprahyoid muscles during different lingual exercises. Audiol Commun. 2015;20(3):203–9.
- 31. Vaiman M, Eviatar E, Segal S. Surface electromyographic studies of swallowing in normal subjects: A review of 440 adults. Report 2. Quantitative data: Amplitude measures. Otolaryngology Head and Neck Surgery. 2004;131(5):773–80.
- 32. Oommen ER. Effects of Three Lingual Conditions on Submental Muscle Activity in Healthy Young and Old Adults. Ohio University; 2013.
- 33. Rogus-Pulia N, Rusche N, Hind JA, Zielinski J, Gangnon R, Safdar N, et al. Effects of device-facilitated isometric progressive resistance oropharyngeal therapy on swallowing and health-related outcomes in older adults with dysphagia. J Am Geriatr Soc. 2016;64(2):417–24.
- 34. Steele CM, Bayley MT, Peladeau-Pigeon M, Nagy A, Namasivayam AM, Stokely SL, et al. A Randomized Trial Comparing Two Tongue-Pressure Resistance Training Protocols for Post-Stroke Dysphagia. Dysphagia. 2016;31(3):452–61.
- 35. Bingjie L, Tong Z, Xinting S, Jianmin X, Guijun J. Quantitative videofluoroscopic analysis of penetration-aspiration in post-stroke patients. Neurol India. 2010;58(1):42–7.
- 36. Zhang Z, Perera S, Donohue C, Kurosu A, Mahoney AS, Coyle JL, et al. The Prediction of Risk of Penetration–Aspiration Via Hyoid Bone Displacement Features. Dysphagia. 2020;35(1):66–72.
- 37. Hughes TD. The Effect of Two Rehabilitation Exercise on Submental Hyolaringeal Muscular Activity. Texas Christian University; 2015.
- 38. Steele CM, Bailey GL, Chau T, Molfenter SM, Oshalla M, Waito AA, et al. The relationship between hyoid and laryngeal displacement and swallowing impairment. Clin Otolaryngol. 2011;36(1):477–9.
- 39. Han H, Shin G, Jun A, Park T, Ko D, Choi E, et al. The relation between the presence of aspiration or penetration and the clinical indicators of dysphagia in poststroke survivors. Ann Rehabil Med. 2016;40(1):88–94.
- 40. Pearson WG, Hindson DF, Langmore SE, Zumwalt AC. Evaluating swallowing muscles essential for hyolaryngeal elevation by using muscle functional magnetic resonance imaging. Int J Radiat Oncol Biol Phys. 2013;85(3):735–40.
- 41. Kim H, Kown Y, Choi H. Home Based Dysphagia Rehabilitation for Stroke Patients Using Information and Communication Technology. J Int Acad Phys Ther Res. 2021;12(1):2267–71.
- 42. Bingjie L, Tong Z, Xinting S, Jianmin X, Guijun J. Quantitative videofluoroscopic analysis of penetration-aspiration in post-stroke patients. Neurol India. 2010;58(1):42–7.
- 43. Zhang Z, Perera S, Donohue C, Kurosu A, Mahoney AS, Coyle JL, et al. The Prediction of Risk of Penetration—Aspiration Via Hyoid Bone Displacement Features. Dysphagia

[Internet]. 2020;35(1):66-72. Available from: https://doi.org/10.1007/s00455-019-10000-5

**Table 3.** Comparison of Parameters Before and After Training in the Intervention and Control Groups

| Parameter | | Group | Baseline | Week 8 | p-value |
|---|---|---|---|---|---|
| Anterior hyoid movement (%C2–C4) | | Intervention | 15.75 (3.21–24.43) | 28.26 (3.5–45.18) | $0.038^{w}$ |
| | | Control | 14.09 (0.96–17.54) | 14.48 (1.07–23.69) | $0.161^{\text{w}}$ |
| | | p-value between groups | $0.178^{\rm m}$ | 0.021 <sup>m</sup> | |
| Superior hyoid mo | vement (%C2–C4) | Intervention | 14.52 (5.54–38.85) | 22.07 (4.83–38.33) | $0.086^{w}$ |
| | | Control | 16.56 (10.68–34.62) | 19.50 (1.77–48.93) | $0.327^{\mathrm{w}}$ |
| | | p-value between groups | $0.441^{\rm m}$ | $0.564^{\rm m}$ | |
| PTT (seconds) | | Intervention | 0.63 (0.1–1) | 0.73 (0.23–0.83) | 0.859 <sup>w</sup> |
| | | Control | 0.68 (0.5–1) | 0.74 (0.33–5.6) | $0.327^{\mathrm{w}}$ |
| | | p-value between groups | $0.923^{\rm m}$ | $0.310^{m}$ | |
| PAS | | Intervention | 4 (2–8) | 2 (1–8) | $0.232^{w}$ |
| | | Control | 4.5 (2–8) | 2 (1–8) | $0.753^{w}$ |
| | | p-value between groups | $1.000^{\rm m}$ | $0.797^{\rm m}$ | |
| m) | Mann-Whitney | Test; | w) | Wilcox | con |